CLINICAL TRIAL: NCT02887573
Title: Free-residue Nutrients for the Bowel Preparation of Colon Capsule Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaichun Wu (Other)
Responsible Party: Sponsor-Investigator, Kaichun Wu, President of Xijing Hospital of Digestive Diseases, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XijingHDD
Record Dates: First submitted 2016-08-20; First posted 2016-09-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Colorectal Polyps
Keywords: Bowel preparation; Colorectal polyps; Colon capsule endoscopy
MeSH Terms: interventions — Endoscopy; Polyethylene Glycols; mosapride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Free-residue nutrients+PEG (Experimental): Diet: Free-residue nutrients Free-residue nutrient will be given when the patients are hungry before the two days of the capsule day.There are no other diet in this arm.
  Drug: PEG 2L PEG are used at 05:00-07:00 the morning of the test. Drug: Mosapride citrate The patients will take 5mg mosapride citrate at 8:00. Drug:PEG 0.75L and 0.50L PEG are administered as boosters for patients. Procedure: Colon capsule endoscopy The colon capsule will be ingested at 08:30 the day of the test.The images will be reviewed by two experienced endoscopists.
  Procedure: Colonoscopy On the following day of the test.All participants will undergo therapeutic colonoscopy.
  Interventions: Drug: Free-residue nutrients; Procedure: Colon capsule endoscopy; Drug: 2L PEG; Drug: PEG; Drug: Mosapride citrate
- Low fiber diet+PEG (Experimental): Diet: Low fiber diet Before the two days of the capsule day,when the patients hungry,low fiber diet wiil be given.
  Drug: PEG 4L PEG are used at 21:00-23:00 the night before the test and 05:00-07:00 the morning of the test.
  Drug: Mosapride citrate The patients will take 5mg mosapride citrate at 8:00. Drug:PEG 0.75L and 0.50L PEG are administered as boosters for patients. Procedure: Colon capsule endoscopy The colon capsule will be ingested at 08:30 the day of the test.The images will be reviewed by two experienced endoscopists.
  Procedure: Colonoscopy On the following day of the test,All participants will undergo therapeutic colonoscopy.
  Interventions: Drug: Low fiber diet; Procedure: Colon capsule endoscopy; Drug: 4L PEG; Drug: PEG; Drug: Mosapride citrate

INTERVENTIONS:
Drug: Free-residue nutrients — This trial evaluated the efficiency of free-residue nutrients for the bowel prepartion of CCE.
  Arms: Free-residue nutrients+PEG
Drug: Low fiber diet — Low fiber diet often used in the bowel prepartion of CCE. In this study, it is the control group.
  Arms: Low fiber diet+PEG
Procedure: Colon capsule endoscopy — In the study,all patients should undergo two colonoscopies.The first is for examinations and the second for therapy.
Drug: 2L PEG — 2L PEG are laxatives for experiment group.
  Other Names: polyethylene glycol
  Arms: Free-residue nutrients+PEG
Drug: 4L PEG — 4L PEG are laxatives in the control group.
  Other Names: polyethylene glycol
  Arms: Low fiber diet+PEG
Drug: PEG — These PEG are for boosters. All patients will take 0.75L and 0.5L PEG for two boosters.
  Other Names: polyethylene glycol
Drug: Mosapride citrate — 5mg mosapride citrate are used to promote gastric motivity.

SUMMARY:
Colon capsule endoscopy(CCE) is a new diagnostic method of colonic lesions.It has advantages of no requirement for sedation and air insufflation.The bowel preparation has a closely relationship with yield of diagnosing diseases.Bowel preparation of CCE is not only to clean the colon but also to promote capsule propulsion.Now there is not an optimal method for CCE.

DETAILED DESCRIPTION:
Objective: In this study, a new bowel preparation regime of the colon capsule is used.This regime combines free-residue nutrients and polyethylene glycol (PEG) to achieve a better preparation quality.

Methods: Participants who underwent a diagnostic colonoscopy examination that demonstrated a colorectal polyps that required endoscopic treatment will be recruited to patients in the study. The first 32 participants receive a traditional low fiber diet two days before the test.Then the patients will take 2L polyethylene glycol (PEG) at 21:00-23:00 before the test day and 2L PEG at 05:00-07:00 on the test day for bowel preparation. The subsequent 30 participants receive two-days free-residue nutrients without other diet before the test.Then the patients will take 2L PEG at 05:00-07:00 on the examination day for bowel preparation. Then they will take 5mg mosapride citrate at 8:00 and ingest the colon capsule at 8:30.0.75L and 0.50L PEG are administered as boosters.And the therapeutic endoscopy will be given on the following day.Before the therapeutic colonoscopy, the participants will take 2L PEG. The colon capsule results will be reviewed by two experienced endoscopists who are blinded to first endoscopy results.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age.
* underwent a diagnostic OC that demonstrated colorectal polyps that required endoscopic treatment.

Exclusion Criteria:

1. dysphagia/swallowing disorder
2. prior major abdominal surgery of the gastrointestinal tract, known or suspected bowel obstruction
3. cardiac pacemaker/implanted electromedical device
4. pregnant or nursing women
5. any allergy or contraindication to the drugs used in the study.
6. refused to sign a informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Bowel Cleansing Level of Two Different Bowel Preparation Methods | an expected average of 1 months from study procedure
  The first 32 patients adopted a low fiber diet two days before the CCE procedure. Bowel preparation included the ingestion of 2L polyethyleneglycol in the evening before test day and 2L PEG in the morning on the test day. The subsequent 30 patients were received free-residue Nutrients。Then they ingested 2L PEG between 5:00 and 7.00 am of the examination day. The capsule was scheduled at 8:30 am. When the capsule reached the small bowel, 0.75L PEG was used as first booster. If the capsule had not been excreted 3 hours later, the patients was received 0.5L PEG.

SECONDARY OUTCOMES:
Accuracy parameters:assessment the yield of detection of polyps ≥6mm and ≥10mm; | an expected average of 1 months from study procedure
The gastrointestinal tract transit times and the colonic transit times between two different bowel preparation methods for CCE; | an expected average of 1 months from study procedure
  The gastrointestinal tract transit time was defined as the time from initial ingestion to capsule excretion. The colon transit time defined as first capsule image of the cecum to capsule excretion.
Colon capsule excretion rate between two different bowel preparation methods; | an expected average of 1 months from study procedure
Adverse events between two different bowel preparation methods. | the PillCam procedure day

CONTACTS AND LOCATIONS:
Overall Officials: Wu Kaichun, phD, Study Director — Xijing Hospital of Digestive Diseases

IPD SHARING:
Plan to Share IPD: Undecided